CLINICAL TRIAL: NCT05729347
Title: Treatment of Parental Anxiety With Virtual Reality (VR): A Prospective, Randomized Study
Brief Title: Treatment of Parental Anxiety Virtual Reality (VR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69068
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Parents; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants will be immersed in a virtual environment. Calming scenery will be shown via the headset for 20-30 minutes
  Interventions: Behavioral: Virtual Reality headset with calming scenery
- Control (No Intervention): No intervention (i.e. virtual reality headset) will be applied to the participant.

INTERVENTIONS:
Behavioral: Virtual Reality headset with calming scenery — Participants will be immersed in a virtual environment. Calming scenery will be shown via the headset for 20-30 minutes
  Arms: Virtual Reality

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headset) are more effective than the standard of care (i.e., no technology based distraction) for preventing anxiety in parental and pediatric populations

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-99 (Parents whose children is hospitalized)
* Able to consent
* Parents whose child is undergoing various procedures at LPCH and Stanford Hospital and Clinics.

Exclusion Criteria:

* People who do not consent
* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Current Nausea
* Seizures
* Visual Problems
* Patients whose children are clinically unstable or require urgent/emergent intervention

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | immediately after the intervention
  Anxiety level measured by a Visual Analogue Scale - Anxiety (VAS-A) ranging from 0-10. Scale ranges from 0-10, with higher scores indicating higher anxiety levels.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | baseline, immediately after the intervention
  The State-Trait Anxiety Inventory (STAI) is a validated self-report questionnaire consisting of two subscales that measure state anxiety (temporary condition) and trait anxiety (general tendency). Each subscale contains 20 items rated on a 4-point Likert scale. Scores range from 20 to 80 per subscale, with higher scores indicating greater anxiety.
Modified Pain Catastrophizing Scale | immediately after intervention
  Modified Pain Catastrophizing Scale(PCS); It is a self-report measure adapted from the Adult Pain Catastrophizing Scale used to assess negative thinking associated with pain. It contains 3 items rated on a 5-point scale ranging from 0 = "not at all" to 4 = "very much".
Device satisfaction | immediately after intervention
  To evaluate the overall impact of device satisfaction, participants will complete the self-developed satisfaction survey. Participants will rank each factor on a Likert scale from 1 = not at all to 5 = a lot.
Procedural-Related Anxiety | Duration of intervention, approximately 20-30 minutes
  Validated questionnaires regarding anxiety will be administers pre- and post-intervention (i.e virtual reality) and compared to those in the control arm (i.e no virtual reality)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang ZY, Kang GC, Koh EYL, Fong RJK, Tang J, Goh CK, Tan NC. Immersive Virtual Reality in Alleviating Pain and Anxiety in Children During Immunization in Primary Care: A Pilot Randomized Controlled Trial. Front Pediatr. 2022 Mar 25;10:847257. doi: 10.3389/fped.2022.847257. eCollection 2022. PMID 35402359